CLINICAL TRIAL: NCT04893564
Title: Prognostic Value of Circulating Tumoral DNA After the First 6 Months of Treatment in Patients With Waldenström Macroglobulinemia
Acronym: SLP-rares
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Henri Becquerel (Other); University Hospital, Caen (Other); University Hospital, Lille (Other); Centre Hospitalier de Lens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2019_843_0024
Record Dates: First submitted 2021-05-17; First posted 2021-05-19 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Waldenstrom's Disease; Waldenstrom Macroglobulinemia
Keywords: Waldenstrom's Disease; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Biological: bone marrow sample — 8 to 13 ml bone marrow sample for frozen storage within one of the 5 certified biobank of the canceropole area.
Biological: blood sample — 20 ml blood sample for frozen storage within one of the 5 certified biobank of the canceropole area.

SUMMARY:
Waldenström Macroglobulinemia (WM) is defined by a bone marrow lymphoplasmacytic infiltration and the presence of a monoclonal immunoglobulin M (IgM) in blood. This chronic lymphoproliferative disorder requires treatment only in case of symptoms, according to accurate criteria described during the second Workshop on WM i.e. in case of cytopenia, bulky organomegaly, immunological or physicochemical consequences of the presence of IgM in circulating blood. A MYD88 mutation, typically a MYD88(L265P), is found in 90% of WM patients. Other gene abnormalities have been observed, the most frequent is a mutation in the CXCR4 gene. Overall, gene mutations in WM involve only a limited number of signalling pathways, yielding the activation of NFkB, namely : the TLR and MYD88 pathway (with an activation of NFkB and BTK in case of MYD88(L265P) mutation), the BCR pathway (involving btk and associated with activations of both NFkB, and erk akt pathway) and the CXCR4 pathway (CXCR4 is a receptor of CXCL12, it is also associated with activations of ERK/MAPK and PI3K). Abnormalities of some of genes, such as TP53, of the expression of the protein CXCL13 and genes involved in the interleukin 6 secretion have been associated with some clinical characteristics.

The purpose of this project is to define the prognostic role of the detection of circulating tumoral DNA (ctDNA) at the end of treatment for the progression/relapse risk within the first 3 years after the first 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient with WM according to diagnostic criteria
* Patients with WM followed in one of the centre of North-Western region.
* Patients requiring first-line or subsequent-line therapy
* Patients agreement for giving informed consent.
* Social insurance system affiliation

Exclusion Criteria:

* Patients with another chronic B-cell malignancy
* patients with other lymphoplasmacytic proliferations
* patients with marginal zone lymphoma.
* Patients with WM and histologic transformation
* Absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
association between circulating tumoral DNA detection and progression-free survival | 3 years
  To define the prognostic role of the detection of circulating tumoral DNA (ctDNA) at the end of treatment for the progression/relapse risk within the first 3 years after the first 6 months of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No